CLINICAL TRIAL: NCT01991886
Title: A Pilot Study to Determine the Feasibility of the Use of Nasal High Flow From Birth in Premature Infants Born at Less Than or Equal to 30 Week Gestational Age.
Brief Title: Using Nasal High Flow From Birth in Premature Infants - a Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ashford and St. Peter's Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2013PR01; 131594 (Other: IRAS)
Record Dates: First submitted 2013-11-11; First posted 2013-11-25 (Estimated); Last update posted 2016-08-12 (Estimated); Status verified 2016-08

CONDITIONS: Premature Birth
Keywords: nasal High Flow; premature baby; CPAP (Continuous positive airways pressure)
MeSH Terms: conditions — Premature Birth; Microcephaly, Primary Autosomal Recessive, 6

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- nasal High Flow applied (Experimental): Application of nasal High Flow 6-7l/min via nasal prongs after birth using a mobile Vapotherm Precision Flow device
  Interventions: Device: Vapotherm Precision Flow

INTERVENTIONS:
Device: Vapotherm Precision Flow — Application of nasal High Flow using 6-7 l/min delivered by nasal prongs from birth
  Other Names: nasal High Flow device; nasal heated humidified high flow cannula

SUMMARY:
Recent large studies have shown that not all premature babies need to be intubated (have a breathing tube inserted) and ventilated, nor do they all need to be given lung surfactant routinely. Those studies showed that even very small babies can be safely supported using nasal Continuous Positive Airway Pressure (nCPAP) which is applied tightly to the nose using nasal prongs. This is a type of noninvasive ventilation (NIV) so that the babies continue to breath, albeit with additional support to reduce their work of breathing. However nCPAP has some drawbacks, including that it can cause skin damage to the nose, and that the heating and humidification of the gas is not always sufficient. We have been using, for over 5 years, a different system to support babies after routine intubation. This is another type of noninvasive ventilation called nasal High Flow (nHF) for which we use a Vapotherm Precision Flow device. Published trials show that it is at least as effective as nCPAP to provide NIV and to prevent the subsequent need for intubation and/or surfactant. However nHF is superior to nCPAP in respect it does not cause nose damage and its heating and humidification is excellent. This pilot study aims to describe and evaluate the use of nHF, using a standard commercially available system (Precision Flow, Vapotherm Inc.), from birth, in babies born less than 30 completed weeks gestation, with a view to avoiding intubation and ventilation. This study is important to establish the feasibility of using nHF immediately after birth.

DETAILED DESCRIPTION:
We propose to pilot the use of this mobile nHF unit, using the Vapotherm Precision Flow device, in the premature population of babies who would normally be either intubated and given surfactant routinely, or be maintained on nCPAP until arrival on the Neonatal Intensive Care Unit (NICU) then transferred onto nHF. Parents will be informed about the pilot and their permission will be sought. We aim to recruit 40 babies less than 30 weeks gestation.

The reason for undertaking a pilot study of this nature is to establish feasibility and proof of concept. It is not designed to be compared to using nCPAP to stabilise babies immediately after birth (although that will be the next and logical progression if this proves to be a feasible technique).

The hypothesis is that using nHF to stabilise babies immediately after birth will confer the same advantages as using nCPAP to stabilise babies in this way, which has been demonstrated in the worldwide literature. For units such as ours who use nHF in preference to nCPAP, this will be an important step in further defining the management of these babies after birth. There is evidence that nHF is at least as good as nCPAP in preventing intubation and reducing lung disease, and it may also offer additional advantages from humidification and reduction in nasal trauma.

The major challenge for this pilot project will be to identify eligible deliveries in a timely manner to ensure that a suitable member of staff is available to speak to parents and gain consent.

Once a delivery has been identified and the parents have agreed to take part, then the following process will take place to manage the newborn baby.

Check the mobile nHF unit

* The mobile nHF unit should be kept plugged in so that the uninterruptable power supply (UPS) is fully charged
* To use it, unplug it to check that the UPS is functioning (green lights indicate full charge), set up a Vapotherm circuit(as per normal routine) and start the machine running on UPS power supply.
* Gas supply should be from the cylinders to check that the pressures are 50bar in both air and oxygen cylinders
* Set the temperature to 37 degrees Celsius
* Once running, turn the unit off if not immediately needed or plug into the mains power and gas(es) where available to conserve gas. The unit can be run on a flow of 1 litre/minute whilst "ticking over" to conserve cylinder gas if needed.
* The prongs should be attached to the circuit.

Once the baby is born

* Place the baby in a polythene bag (as per normal practice)
* Ensure the baby is breathing. If not, or the baby is bradycardic, then normal resuscitation measures should be applied. It will only be appropriate to apply the mobile nHF if the baby is breathing and is clinically stable.
* Once the baby is born, increase the flow to 6 litres/min
* If the baby is breathing then apply the nHF prongs and observe carefully
* Suction should only be applied gently, if needed to remove excessive secretions in the mouth and throat. Babies on high flow will often "blow bubbles" and there may be lung fluid in the throat, but suction should not be vigorous
* Apply a saturation monitor (as per normal practice) to check Heart Rate (HR) and Oxygen Saturation (SaO2).
* Dry the baby's face sufficiently to be able to apply duoderm dressing to stick down the prongs to the cheeks.
* Observe the baby carefully, ensure attention to thermal care and inform the parents about progress.
* As soon as the baby appears stable, move to NICU as per normal practice

Transfer to NICU

* Two people are needed to effect the transfer from labour ward/theatre to NICU, one to move the mobile nHF and one to move the resuscitaire.
* On arrival in NICU, plug the mobile nHF into gas and power supplies (switch the manifold over)
* Ensure that there is a second, cotside Vapotherm (empty) unit
* Leave the baby in the resuscitaire and check the admission temperature.
* Stop the mobile nHF, remove the cartridge and place it into the cotside Vapotherm unit. Start it running, it should run straight away. Ensure that the correct temperature, flow and Fraction Of Inspired Oxygen (FiO2) are set
* This process takes less than 20 seconds and as the baby is breathing will not be detrimental
* Transfer the baby into the incubator and commence normal admission practices
* Document the resuscitation clearly in the baby's notes

Cleaning and charging the mobile nHF

o Remove the mobile nHF, clean the Vapotherm Precision flow nHF unit. Ensure the cylinders are switched off and plug into the wall to recharge the UPS.

ELIGIBILITY:
Inclusion Criteria:

* Parental consent
* 24+0 to 30+0 weeks(agreed dates) gestation born alive
* Breathing spontaneously at birth or soon after with minimal resuscitation
* Oxygen saturations >90% by 5 minutes

Exclusion Criteria:

* No parental consent
* Born in poor condition and unlikely to survive
* Needing resuscitation including intubation and/or chest compressions
* Not breathing and thus needing intubation
* Oxygen saturations <90% by 5 minutes
* <24 weeks gestation
* >30 weeks gestation

Ages: 24 Weeks to 30 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 28 (Actual)
Dates: Start 2014-01; Primary Completion 2015-01 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Need for endotracheal intubation prior to admission to Neonatal Unit | From birth
  Babies who are clinically stable will not require intubation prior to admission to the neonatal unit.

SECONDARY OUTCOMES:
Development of pneumothorax within 24 hours of birth | First 24 hours after birth
  Pneumothorax is a rare but important outcome measure.
Requirement for endotracheal intubation and surfactant administration after admission to neonatal unit within 24 hours of birth | First 24 hours after admission to neonatal unit
  Intubation and surfactant administration after admission within the first 24 hours indicates severe respiratory distress syndrome requiring treatment according to agreed local protocols
Development of bronchopulmonary dysplasia defined as oxygen requirement at 36 weeks corrected age | Defined at 36 weeks corrected age
  Bronchopulmonary dyplasia is an important outcome of the respiratory management of premature babies. We use the standard definition of an ongoing oxygen requirement at 36 weeks corrected age with compatible X-ray changes.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Dr Reynolds, PhD, Principal Investigator — Ashford and St. Peter's Hospitals NHS Foundation Trust
Locations (1):
- Neonatal ICU, St Peter's Hospital, Chertsey, Surrey, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Reynolds P, Leontiadi S, Lawson T, Otunla T, Ejiwumi O, Holland N. Stabilisation of premature infants in the delivery room with nasal high flow. Arch Dis Child Fetal Neonatal Ed. 2016 Jul;101(4):F284-7. doi: 10.1136/archdischild-2015-309442. Epub 2016 Jan 5. PMID 26733541